CLINICAL TRIAL: NCT05347186
Title: Effects of 8-weeks Systematic Corrective Exercise Program on Body Posture and Stability in Pronation Distortion Syndrome
Brief Title: Effects of 8-weeks Systematic Corrective Exercise Program in Pronation Distortion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0132 Ghazal Hussain
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Pronation; Ankle; Distortion
Keywords: Pronation; Posture; Distortion; Navicular; Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic corrective exercises and non-biomechanical functional exercises (Experimental)
  Interventions: Other: Systematic corrective exercises and non-biomechanical functional exercises; Other: Non biomechanical functional exercises
- Non biomechanical functional exercises. (Other)
  Interventions: Other: Non biomechanical functional exercises

INTERVENTIONS:
Other: Systematic corrective exercises and non-biomechanical functional exercises — 1. Restraint exercise or self-release: will involve the gastrocnemius muscle, soleus muscle, fibula, knee compressor muscles, adductors of the thighs, the short head of the biceps femoris, and iliotibial band for 30 seconds, using a foam roller.
  2. Static stretching drills: involving the soleus and gastrocnemius muscles on an inclined plane, tensor fasciae latae muscle, short head of the biceps femoris, and ilio- psoas muscle;
  3. Resistance exercises: will consist of strengthening the eccentric muscles of the feet including dorsiflexion and knee inversion, adduction, and extension, external rotation of the hip joint with TheraBand exercise band, and strengthening the intrinsic muscles of the foot.
  4. Integrative exercises: including the star balance test on all planes and resistive exercises.
  Arms: Systematic corrective exercises and non-biomechanical functional exercises
Other: Non biomechanical functional exercises — Conventional treatment involved Non biomechanical Functional exercises (NBF), these exercises indicated for the control group consists of dorsal and plantar flexion of the metatarsophalangeal joints in unloading of the subject in a long sitting position on a chair or couch with the knee at 90◦ for a period of eight weeks. Feet will be in hanging position to allow plantar flexion smoothly. The exercises will carry out daily without any kind of resistance for a period of 30s. A total of five series will be completed for each foot. These exercises will be considered as non-therapeutic which might have affected the foot's posture.

SUMMARY:
Pronation distortion syndrome is a postural complexity of lower extremity which primarily involves hyper pronation of feet leading to other dysfunctional movement patterns throughout the kinetic chain and gait mechanics. Excessive foot pronation is followed by internal tibial rotation and adduction of knees forming knock knees. This lower extremity distortion pattern causes a chain reaction of muscle imbalances. The objective of this study is to determine effects of 8-Weeks Systematic Corrective Exercise program on Body Posture and stability in Pronation Distortion Syndrome. This study will be a Randomized Controlled trial and will be conducted at Riphah college of rehabilitation sciences and Ibrahim medical Centre Lahore. The study will be completed within the time duration of 10 months. Convenient sampling technique will be used to collect the data. A sample size of Total 36 patients will be taken in this study. Patients will be divided into two groups. Group A will be treated with conventional treatment along with systematic corrective exercise program. Group B will be given conventional treatment only. The groups will participate in the training program one day after the pre-test, three sessions per week for two months. The diagnosis of pronation distortion will be detected by navicular drop in detectable flat feet without pain. Variables to be tested will be, functional movement screen test, navicular drop, knock knees and lordosis, and will be measured before the start of treatment and after 8 weeks of treatment. Data will be analyzed on SPSS 25.

DETAILED DESCRIPTION:
Pronation distortion syndrome is a common postural distortion of the lower extremity, involving the anterior part of the leg. In this deformity, the head of the talus and navicular bones are rotated inward and downward, and the body's center of gravity shifts inward, resulting in flat feet. It may cause pain in the leg and disturbances in the tarsal part, in addition to distal and proximal parts. Excessive foot pronation include inward rotation of the tibia, internal rotation of the thighs associated with flat feet, genu valgum (knock-knee), and increased lordosis thus causing abnormalities in lumbo-pelvic region and lower limb.

In this deformity, peroneal muscle, gastrocnemius muscle, hamstrings, soleus muscle, iliotibial band, adductors, and psoas muscle are functionally tightened, while posterior and anterior tibialis, gluteus Medius, gluteus maximus, vastus medialis, and hip external rotators are inhibited. Excessive pronation will misalign the entire lower body, reducing the ability of powerful muscles like the quadriceps and glutes to maintain force production. Length tension relationships establish that the resting length of a muscle determines whether it can generate optimal tension, if the feet excessively flatten and the femur excessively rotates and adducts, then the joints don't stack, the tissues don't load, and energy is lost. Over time, tissues may become irritated, inflamed or even weakened, which often leads to more serious problems, such as ruptured tendons or stress fractures . The body weight normally falls on the center of the foot, and balance is maintained by the muscle activity of the foot. If the foot becomes diseased or deformed, the foot adapts to perform its functions under the conditions of disease or deformity. Several factors of pronation distortion can increase the likelihood of cuboid syndrome including midtarsal instability, excessive body weight, ill-fitting or poorly constructed orthoses or shoes and inadequate exercise recovery. The postural defects cause pronated subtalar joint, inverted forefoot and instability of mid tarsal joint leading to improper dynamic stabilization. Every degree of subtalar pronation that occurs produces an exponential increase in midtarsal joint instability. Pronated feet are very common among people with flexible flat feet in which the medial longitudinal arch of the foot largely collapses during the stance phase of gait causing over supination and over pronation but restores after removal of body weight. Kinetic coupling of 4 pronated feet alters during improper gait mechanics and results in changes of inter joint angle coordination. This disturbs the inter joint coordination which is involved in determining movement flexibility and stability thus effecting gait pattern leading towards occurrence of injury. In the case of postural distortion, instability and damage to the lower extremity cause hypermobility, and passive instability and more neurological control by the neuromuscular system is required to maintain stability and balance. The instability resulting from a flat foot could cause patho-mechanical problems as well as a compensating action in the close kinematic chain of the lower extremity. Excessive pronation transmitted to internal rotation of the tibia, may cause overloading of the knee joint or may be the cause of other changes in proximal part of the lower extremity. The feet support the body's weight and play the role of levers when an individual is performing work. By performing closed kinetic chain exercises under loads and by increasing the strength of the muscles proximal to the lower extremities, one can correct the hyper pronation of the foot in the distal lower extremities and can prevent ligamentous laxity. This study will determine the effects of 8 weeks systematic corrective exercises on body posture and stability in pronation distortion syndrome. PDS is a postural defect that occurs by initiation of foot hyper pronation that further causes forced tibial rotation, knock knees and progression of lumbar lordosis. Studies suggest women are more prone to pronated feet than men recording prevalence of 20-30 percent.

Furthermore, biomechanical abnormalities reported to be prevalent as 60-90 percent.

In 2020 Ali Golchin et al conducted a study to emphasize on the postural deformities caused by pronation distortion syndrome. It was a randomized controlled trial. In this study functional movement screening were performed to evaluate subjects' performance. Treatment protocol included systematic and corrective exercise program that concluded reduction in likelihood of injury and improvement in posture with subjects with pronated feet.

In year 2020 Marina gil-calvo et al studied the effects of custom-made and prefabricated foot orthoses on kinematic parameters in recreational runners with flat feet dysfunction.

Initial field test was monitored to determine individuals maximum aerobic speed in athletes.

Subjects with history of foot orthosis implementation were excluded. There were three groups, one with custom orthosis, 2nd group underwent with prefabricated orthosis and 3 rd was control group. Foot eversion parameters were measured before and after the intervention.

Findings of the study suggested no significant difference in improvement even after weeks of intervention. Modification in the running mechanics to maintain ideal movement pattern in runners were suggested for better outcome . In 2020 Manuel Pabón-Carrasco et al checked the association of short foot exercises (SFE) with Non biomechanical function (NBF) exercises in the strength development of intrinsic muscles of pronated feet. The intrinsic foot muscle is considered primordial in maintaining the plantar arch and controlling foot posture. A randomized clinical trial was carried out with 85 asymptomatic participants with a bilateral Foot Posture Index (FPI) greater than 6 points.

The pronation of each foot were measured twice. Changes were observed in the ND and FPI pre-intervention and post-intervention for the subjects of each independent group. A tendency of a more neutral position and a decrease of the ND were noted. 6 In 2019, according to Nikkhouamiri F et al, postural abnormalities due to dysfunction of pronated feet can irritate the functional and balance kinematic of walking resulting in skeletal abnormalities and postural control disorder. Navicular drop test was used to asses the flat feet deformity. Given the results, application of corrective exercise program on improving balance and function in female population were effective. Female adolescents showed improved postural control, coordination and stability. Farhan Alam et al in 2019, worked on selective strengthening of tibialis posterior and stretching of iliopsoas on navicular drop, dynamic balance, and lower limb muscle activity in pronated feet. A previous study reported that 20% of the adult population have flatfeet and 12.8% of adults with flatfeet are males and 14.4% are females. The experimental group performed stretching and strengthening of tibialis anterior, iliopsoas and adductor muscles whereas conventional group performed towel curl exercises. Improvement in biomechanical alignment was noted in this study. Ru-Lan Hsieh, MD et al in 2018, conducted a randomized controlled trial study to measure the effects of customized arch support insoles in children with flexible flat and pronated feet.

In this 12-week intervention program subjects went through the measurement of calcaneal inclination angle; hypermobility score and navicular drop test. Physical activity i.e., 10-m normal and fast walking, stair ascent, stair descent, and chair rising were assessed within the intervention. The insoles helped subtalar joint to maintain its normal neutral position during mobility (14). The literature suggests to conduct a study on both males and females with age group more than 16 years. There has been studies that has worked on foot for correction of pronation but the correction of kinetic chain disturbance due to hyper pronation has been in neglection. Given the prevalence of flat feet and influence of proximal and distal chains, this study will be conducted to determine effects of 8-Weeks Systematic CCorrective Exercise program on Body Posture and stability in Pronation Distortion Syndrome.

ELIGIBILITY:
Inclusion Criteria:

Age 18-25 years

* Male and female university going students
* Navicular drop test greater than 10mm .
* Detection of flexible flat feet without pain.
* Having a normal vision or corrected vision using spectacles or contact lenses

Exclusion Criteria:

The presence of pain or emergence of pain during the study.

* Congenital abnormalities such as club foot, common peroneal nerve injury.
* Visible deformation of foot.
* History of surgery on the ankle, knee, thighs, hip, or back
* Use of assisted devices while walking

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Functional Movement screen test | 8 weeks
  The Functional Movement Screen (FMS) test has been used for devising functional evaluation programs. This set of tests was designed using 7 movement patterns for the simultaneous evaluation of mobility and stability. This set of tests include the deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up, and rotatory stability. The intrarater test-retest and interrater reliability of the FMS composite score resulted in an ICC of 0.76
Navicular drop test | 8 weeks
  It is a simple test that is clinically used to measure the range of eversion and sagittal deformation of the mid-foot.
Valgus angle by Goniometer | 8 weeks
  This factor is determined by measuring the hindfoot valgus angle (the angle behind the ankle).The natural angle is 180 and an angle more than 9 degrees is considered as hyper pronation. Ankle dorsiflexion reliability, ICC 0.12-0.73 and validity 0.51-0.83
Knock Knee by Sliding caliper | 8 weeks
  To measure the distance, the intercondylar and intermalleolar points are identified. The internal condyles of the knee and the protruding parts in the internal area of the lower end of the tibia and the upper section of the ankle joint are considered as the internal ankles of the feet. Then, these distances are measured using a caliper. The intra-rater and inter-rater reliability values of this test have been reported as good and excellent i.e., 0.997
Lumbar lordosis measured by Kidoz Flexible ruler | 8 weeks
  Using this method, the average lordosis angle in healthy individuals is shown to be up to 50.9 degrees and for the age group of younger than 14 years, the angle is up to 34.45 degrees, while for the age group of 15-25 years, the angle up to 32.20 degrees is considered normal.
  Flexible ruler shas high intra-rater reliability to be 0.991

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Ibrahim medical Centre Lahore., Lahore, Punjab Province
  - Riphah Rehabilitation Center, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golchini A, Rahnama N, Lotfi-Foroushani M. Effect of Systematic Corrective Exercises on the Static and Dynamic Balance of Patients with Pronation Distortion Syndrome: A Randomized Controlled Clinical Trial Study. Int J Prev Med. 2021 Oct 19;12:129. doi: 10.4103/ijpvm.IJPVM_303_19. eCollection 2021. PMID 34912505
- [Background] Jafarnezhadgero A, Mousavi SH, Madadi-Shad M, Hijmans JM. Quantifying lower limb inter-joint coordination and coordination variability after four-month wearing arch support foot orthoses in children with flexible flat feet. Hum Mov Sci. 2020 Apr;70:102593. doi: 10.1016/j.humov.2020.102593. Epub 2020 Feb 28. PMID 32217211
- [Background] Goo YM, Kim TH, Lim JY. The effects of gluteus maximus and abductor hallucis strengthening exercises for four weeks on navicular drop and lower extremity muscle activity during gait with flatfoot. J Phys Ther Sci. 2016 Mar;28(3):911-5. doi: 10.1589/jpts.28.911. Epub 2016 Mar 31. PMID 27134383
- [Background] Gil-Calvo M, Jimenez-Perez I, Priego-Quesada JI, Lucas-Cuevas AG, Perez-Soriano P. Effect of custom-made and prefabricated foot orthoses on kinematic parameters during an intense prolonged run. PLoS One. 2020 Mar 26;15(3):e0230877. doi: 10.1371/journal.pone.0230877. eCollection 2020. PMID 32214390
- [Background] Pabon-Carrasco M, Castro-Mendez A, Vilar-Palomo S, Jimenez-Cebrian AM, Garcia-Paya I, Palomo-Toucedo IC. Randomized Clinical Trial: The Effect of Exercise of the Intrinsic Muscle on Foot Pronation. Int J Environ Res Public Health. 2020 Jul 7;17(13):4882. doi: 10.3390/ijerph17134882. PMID 32645830
- [Background] Alam F, Raza S, Moiz JA, Bhati P, Anwer S, Alghadir A. Effects of selective strengthening of tibialis posterior and stretching of iliopsoas on navicular drop, dynamic balance, and lower limb muscle activity in pronated feet: A randomized clinical trial. Phys Sportsmed. 2019 Sep;47(3):301-311. doi: 10.1080/00913847.2018.1553466. Epub 2018 Dec 5. PMID 30517043
- [Background] Haun C, Brown CN, Hannigan K, Johnson ST. The Effects of the Short Foot Exercise on Navicular Drop: A Critically Appraised Topic. J Sport Rehabil. 2020 May 8;30(1):152-157. doi: 10.1123/jsr.2019-0437. PMID 32384261
- [Background] Ore V, Nasic S, Riad J. Lower extremity range of motion and alignment: A reliability and concurrent validity study of goniometric and three-dimensional motion analysis measurement. Heliyon. 2020 Aug 25;6(8):e04713. doi: 10.1016/j.heliyon.2020.e04713. eCollection 2020 Aug. PMID 32904291